CLINICAL TRIAL: NCT01150305
Title: Genetic Epidemiology of Non-syndromic Dominant Deafness
Brief Title: Epidemiology of Non-syndromic Dominant Deafness
Acronym: SURDOM
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AOM 08041
Record Dates: First submitted 2010-03-29; First posted 2010-06-24 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Hearing Impairment
Keywords: Autosomal dominant inheritance; Mutation; Prevalence
MeSH Terms: conditions — Hearing Loss; Multiple Pterygium Syndrome, Autosomal Dominant | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Peripheral whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patient presenting familial dominant non syndromic hearing loss starting between 4 and 40 years old, over 2 generations
  Interventions: Biological: blood sample
- 2: Healthy volunteer from the same families
  Interventions: Biological: blood sample

INTERVENTIONS:
Biological: blood sample — Peripheral whole blood sample, 5 ml

SUMMARY:
Hearing impairment is a common disorder that affects at least 7% of individuals in our countries. Even the causes of hearing impairment are numerous, genetic causes represent the main factor of sensorineural deafness. Among hereditary non-syndromic deafness autosomal-dominant inheritance is observed in about 10-20% of the cases. These forms of deafness are usually post-lingual and progressive. To date more than 41 chromosomal localisation and 21 genes associated to non syndromic dominant deafness have been described. It represents an extreme genetic heterogeneity making difficult the studies of these forms of hearing impairment. But, genetic diagnostic testing is crucial in these cases. Indeed, therapeutic research are in the way to prevent the progression of the disorder. The aim of this work is to establish the prevalence of the different genes involved in these forms of deafness.

DETAILED DESCRIPTION:
The protocol consists first in the recruitment of 150 families with non syndromic dominant hearing impairment. The families will be recruited by the clinical investigators. The clinic and radiological characteristics of the hearing impairment will be collected by the clinical investigators. Samples of patients and healthy relatives will be sent to the referral center. A linkage study of the whole genome by SNP studies is in progress in a cohort of large families affected by autosomal dominant deafness. This work will enable us to select the loci that may be frequently implicated in our population and screen these genes in the 150 families included in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age > 4 years.
* Patient presenting familial dominant non syndromic hearing loss starting between 4 and 40 years old, over 2 generations
* Healthy volunteer from the same families
* Clinical and paraclinical assessment (genetic and ophthalmologic examination, audiometric tests, inner ear CT scan)
* Affiliated to the national health insurance benefit
* Signature of informed consent form

Exclusion Criteria:

* hearing loss resulting from an extrinsic reason or an associated syndrome
* Defective or insufficient samples
* No or insufficient clinical and biological description
* No informed consent form

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: families with non syndromic dominant hearing impairment followed by the clinical investigators
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2009-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
The identification of a deleterious mutation of a gene coding a protein present in the cochlea | 1 day

SECONDARY OUTCOMES:
The phenotype genotype relationships after identification of the causative gene and mutation | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Françoise Denoyelle, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Armand-Trousseau, Service d'ORL pédiatrique et de Chirurgie Maxillo Faciale, Paris, France